CLINICAL TRIAL: NCT07391761
Title: A Multi-center Observational Study of the Effectiveness of Elranatamab in Patients With Relapsed and/or Refractory Multiple Myeloma in Taiwan
Brief Title: A Real World Study of Elranatamab in Patients With RR Multiple Myeloma in Taiwan
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1071049
Record Dates: First submitted 2025-12-15; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Refractory Multiple Myeloma (RRMM)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elranatamab in Patients with Relapsed and/or Refractory Multiple Myeloma: Patients with Relapsed and/or Refractory Multiple Myeloma treated with Elranatamab
  Interventions: Drug: Non intervention

INTERVENTIONS:
Drug: Non intervention — Non intervention

SUMMARY:
The purpose of this study is to evaluate:

* What is the real-world effectiveness of elranatamab in patients with relapsed and/or refractory multiple myeloma (RRMM) in Taiwan?
* What are the baseline and clinical characteristics of RRMM patients who have received eltanatamab in Taiwan?
* What are the treatment patterns of RRMM patients receiving elranatamab in the real-world setting in Taiwan?

DETAILED DESCRIPTION:
This study is seeking participants who:

* have relapsed or refractory multiple myeloma (RRMM),
* have received at least four prior lines of therapy (including a PI, an IMiD, and an anti-CD38 antibody),
* are 18 years or older.

Participants receive elranatamab according to the approved label in Taiwan and continue treatment until disease progression or discontinuation. The study will evaluate real-world effectiveness and describe patient characteristics and treatment patterns to better understand elranatamab use in routine care.

ELIGIBILITY:
Inclusion criteria:

1. Patients age ≥ 18 years at the initiation of elranatamab
2. Patients who have received at least one dose of elranatamab in consistent with the approved label in Taiwan.
3. Evidence of a personally signed and dated informed consent document (ICD) indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study. The ICD waiver is acceptable for patient who was ceased before recruitment.

Exclusion criteria:

Patients who participated in any prior clinical trials using elranatamab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of RRMM patients who have initiated elranatamab in consistent with the local health authority approved product label
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
rwTTR (real-world time to response) | At 1 month, 3 months, 6 months, 9 months, 12 months, and 18 months following initiation of elranatamab treatment (index date.)
  Time from index date to the first documented real-world response.
rwORR (real-world overall response rate) | At 1 month, 3 months, 6 months, 9 months, 12 months, and 18 months following initiation of elranatamab treatment (index date.)
  Proportion of patients achieving real-world overall response at predefined assessment time points.
rwDOR (real-world duration of response） | From first response until 18 months
  Time from the first documented real-world response to real-world disease progression, death, or end of study.
rwPFS (real-world progression-free survival) | From initiation of elranatamab treatment (index date) until 18 months
  Time from index date to the first documented real-world disease progression or death.
rwOS (real world overall survival) | From initiation of elranatamab treatment (index date) until 18 months
  Time from index date to death from any cause.
rwTTNT (real world time to next treatment) | From initiation of elranatamab treatment (index date) until 18 months
  Time from index date to initiation of the next line of anti-myeloma therapy or end of study.

SECONDARY OUTCOMES:
Demographic: Age | At baseline
  Age (measured in years)
Demographic: Sex | From MM diagnosis until index date, and from index date until 18 months
  sex/gender (male/female)
Anthropometric Measures | At baseline
  Height (in cm), weight (in kg), BMI (kg/m²),
ECOG Performance Status | At baseline
  Number and proportion of patients in each ECOG PS category (0-5)
Myeloma-related Clinical Characteristics | At baseline
  Baseline disease characteristics including myeloma type (IgG, non-IgG, light-chain, non-secretory), bone marrow plasma cell %, presence of EMD, ECOG status, CRAB symptoms, ISS/R-ISS stage, MGUS, SMM, and cytogenetic risk.
Laboratory Characteristics | At baseline
  Baseline laboratory result of creatinine clearance (CrCl) categories (stages 1-5 or <30/≥30 mL/min)
Prior Treatment History | At baseline
  Number and proportion of patients with prior ASCT, prior anti-MM therapies
Time from Diagnosis and Line of Elranatamab Treatment | From the index date (initiation of elranatamab treatment) up to 18 months
  Time from MM diagnosis to elranatamab initiation.
Elranatamab Discontinuation and Treatment Modifications | From the index date (initiation of elranatamab treatment) up to 18 months
  Number and proportion of patients with treatment discontinuation (and reasons), dosing or schedule modifications (excluding step-up), and switches from QW to Q2W after 6 cycles.
Subsequent Treatments After Progression | From the index date (initiation of elranatamab treatment) up to 18 months
  Number and proportion of patients receiving subsequent treatments following first progression or discontinuation of elranatamab.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071049